CLINICAL TRIAL: NCT00369174
Title: Phase IIA Trial of Rosiglitazone (Avandia) for Oral Leukoplakia
Brief Title: Rosiglitazone Maleate in Treating Patients With Oral Leukoplakia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2012-02968; 2005-0485; N01CN35159 (NIH); P30CA008748 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-01

CONDITIONS: Oral Leukoplakia
MeSH Terms: conditions — Leukoplakia, Oral | interventions — Rosiglitazone

ARMS (1):
- Treatment (rosiglitazone maleate) (Experimental): Patients receive oral rosiglitazone once daily. Treatment continues for 12 weeks in the absence of unacceptable toxicity.
  Interventions: Drug: rosiglitazone maleate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: rosiglitazone maleate — Given orally
  Other Names: Avandia; BRL49653; ROS
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well rosiglitazone works in preventing oral cancer in patients with oral leukoplakia. Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of rosiglitazone may keep cancer from forming in patients with oral leukoplakia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of clinical response of oral premalignant lesions (OPL) to 12 weeks of therapy with rosiglitazone (Avandia), 8 mg daily, defined as greater than or equal to 50% reduction in the measured product of perpendicular dimension of the target lesion, or improvement in the degree of dysplasia.

SECONDARY OBJECTIVES:

I. To determine the rate and degree of change of putative biomarkers of rosiglitazone efficacy including:

COX-2, cyclin D1, Ki-67, p21/waf1, PPAR gamma, K1 cytokeratin, involucrin, transglutaminase expressions, and TUNEL.

II. To estimate the correlation between DNA ploidy measurements in OPL with clinical response and or response of biomarkers to rosiglitazone therapy, and to estimate the efficacy of rosiglitazone therapy to normalize aberrant DNA ploidy in OPL.

III. To thoroughly assess smoking patterns among trial participants and to examine the relationship of smoking to treatment response.

IV. To assess the safety of this agent in short-term use in this population.

OUTLINE: This is a multicenter, open-label, nonrandomized study.

Patients receive oral rosiglitazone once daily. Treatment continues for 12 weeks in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with a suspected or histologically confirmed index oral premalignant lesion (excluding carcinoma in situ), 12mm or greater in size that has not been biopsied in the past 6 weeks; each index lesion must be either a:

  * dysplastic measurable leukoplakia or erythroplakia in the oral cavity or accessible oropharynx, or
  * hyperplastic leukoplakia of high-risk sites, lateral and ventral tongue and floor of mouth
* The subject's life expectancy is > 12 weeks and Karnofsky performance score is 70-100%
* Hemoglobin and hematocrit levels above the lower limit of normal
* White blood cells >= 3,000/uL
* Platelets >= 125,000/uL
* Total bilirubin =< 1.5 x ULN
* AST (SGOT)/ALT (SGPT) =< 1.5 x ULN
* BUN and serum creatinine =< 1.5 x ULN
* LDH =< 1.5 x ULN
* If the subject is female and of childbearing potential (women are considered not of childbearing potential if they are at least two years postmenopausal and/or surgically sterile), she:

  * has been using adequate contraception (abstinence, IUD, birth control pills, or spermicidal gel with diaphragm or condom) since her last menses and will use adequate contraception during the study, AND
  * is not lactating, AND
  * has a documented negative serum pregnancy test within 14 days prior to randomization
* The subject has discontinued any other oral cancer chemopreventive therapy at least 12 weeks prior to the Baseline visit and all toxicities have been fully resolved; daily aspirin is permitted
* The subject is willing and able to fully participate for the duration of the study
* If applicable, the subject has been counseled on smoking cessation
* The effects of rosiglitazone (Avandia) on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, and because rosiglitazone has been associated with fetal death and growth retardation in rats and rabbits and placental pathology in rats, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately and will be removed from the trial
* Ability to understand and the willingness to sign a written informed consent document
* The subject is of New York Heart Association (NYHA) Class 1 to 4 cardiac status

Exclusion Criteria:

* The subject has active cancer or carcinoma in situ of the head and neck
* The subject has a contraindication to biopsy
* The subject has any history of congestive heart failure, any history of myocardial infarction, angina, or coronary artery disease within the past 6 months, or active cardiac disease
* The subject exhibits clinical evidence of active liver disease, history of chronic liver disease or edema
* The subject currently receives insulin, sulfonylurea or metformin (doses of rosiglitazone greater than 4 mg daily in combination with these therapies are not currently indicated; because this protocol uses the maximum recommended dose of 8 mg daily, subjects on insulin, sulfonylurea or metformin will be ineligible for participation in this trial); the subject is currently receiving thiazolidinediones; the subject is a diabetic not on treatment or hyperglycemic (has a random blood glucose level > 200 mg/dl); the subject has diabetic macular edema
* The subject is currently receiving medical therapy for dysregulated blood sugar
* The subject has experienced jaundice with Rezulin® (troglitazone)
* The subject has known hypersensitivity to rosiglitazone, Avandia, or any of its components
* The subject has a history of colorectal cancer, familial adenomatous polyposis (FAP) or hereditary non-polyposis colorectal cancer (HNPCC)
* The subject has a history of invasive cancer within the past 18 months (excluding non-invasive bladder cancer, non-melanoma skin cancer and in situ cervical cancer); subjects (excluding those with a history of colorectal cancer, FAP or HNPCC) who received curative treatment and have shown no evidence of recurrence for 18 months will be eligible
* The subject has had chemotherapy, immunotherapy, hormonal therapy (other than HRT for menopause), or radiation therapy within 18 months of the Baseline visit
* The subject will need concurrent chemotherapy, radiotherapy, hormonal (other than HRT for menopause), or immunotherapy during the time of study
* The subject has received any investigational medication within 30 days of the Baseline visit or is scheduled to receive an investigational drug during the course of the study
* The subject participated in the study previously and was withdrawn
* The subject is pregnant or nursing
* Subjects who have had the study drug prior to this study
* The subject has uncontrolled intercurrent illness including: ongoing or active infection, HIV, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who show complete or partial response in either clinical or histological outcomes | 12 weeks
  Estimated together with 95% confidence interval. The confidence interval will be constructed using exact binomial confidence intervals (rather than the normal approximation).

SECONDARY OUTCOMES:
Tissue expressions of COX-2, cyclin D1, Ki-67, p21/waf1, PPAR gamma, K1 cytokeratin, involucrin, and transglutaminase, and tissues levels of apoptosis (assessed using TUNEL) | 12 weeks
  Summarized at each time point using summary statistics such as the mean, median, and range. The changes in levels of these biomarkers will also be explored with similar summary statistics and with graphical methods as well.
Tissue DNA ploidy | 12 weeks
Smoking and alcohol use | Up to 12 weeks
  Assessed descriptively. Fisher's exact test may be used to assess whether there is a significant association between smoking status and efficacy of rosiglitazone.
Adverse events defined as any untoward medical occurrence in a study participant, graded using the NCI CTCAE version 3.0 | Up to 12 weeks
  Descriptively summarized in tabular form.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Boyle, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States